CLINICAL TRIAL: NCT01687868
Title: Evaluation of Efficacy and Safety of General Anesthesia Using Dexmedetomidine With Sevoflurane in Patients Undergoing Arthroscopic Shoulder Surgery: Preliminary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2012-0351
Record Dates: First submitted 2012-09-05; First posted 2012-09-19 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Arthroscopic Shoulder Surgery in the Beach-chair Position
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dexmedetomidine continuous infusion (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine 0.7mcg/kg/hr continuous infusion

SUMMARY:
Patients undergoing shoulder arthroscopy in the beach chair position may be at risk for adverse neurologic events due to cerebral ischemia.

Dexmedetomidine, a potent alpha adrenoceptor agonist which dose-dependently reduces arterial blood pressure and heart rate, decreases the hemodynamic and catecholamine response in the perioperative period.

dexmedetomidine has an effect of peripheral vasoconstriction thus it is theologically appropriate for reducing bleeding for arthroscopic operation field.

The aim of this study is to evaluate the efficacy and the safety of dexmedetomidine on cerebral oxygen saturation, cognitive function, hemodynamic stability and operative field in patients undergoing arthroscopic shoulder surgery in the beach-chair position.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Aged between 20 and 70 year
* general anesthesia for arthroscopic shoulder surgery in the beach-chair position

Exclusion Criteria:

* Congestive heart failure, coronary artery occlusive disease
* Bradycardia < 50 BPM, 2nd degree < AV block
* Poorly controlled hypertension
* ß blocker medication
* Coagulopathy
* Pregnancy, nursing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Regional cerebral oxygen saturation value | T1,T2,T3, T4, T5,T6, T7, T8, T9 time of post-dose during surgery
  Before the anesthetic induction(T1), Before endotracheal intubation(T2), After endotracheal intubation(T3), Before the beach-chair position(T4), 5 minutes after the beach-chair position(T5), Before the operation(T6), 5 minutes after the incision(T7), After removal of the arthroscopy(T8), at the end of the operation(T9)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine,Yonsei University Health System, Seoul, Seoul, South Korea